CLINICAL TRIAL: NCT00653692
Title: Methadone, Buprenorphine and Fetal Neurobehavior
Brief Title: Fetal Neurobehavior in Poly-drug Dependent Women
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren M. Jansson, Associate Professor of Pediatrics Johns Hopkins University School of Medicine, National Institute on Drug Abuse (NIDA)
Other Study IDs: 9811; R01DA019934 (NIH); DPMCDA
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Poly Drug Exposed Pregnancies
Keywords: Substance abuse; fetal development; vagal tone
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Poly drug dependent women

SUMMARY:
This project examines fetal neurobehavior and maternal physiology in poly-drug dependent women. This study also evaluates infant neonatal abstinence syndrome, infant neurobehavior and vagal tone in the post-partum period.

DETAILED DESCRIPTION:
Little is known about the link between maternal physiology, fetal neurobehavior and neonatal abstinence syndrome in multiply drug-dependent women. Previous research by this group of investigators has found that the severity of neonatal abstinence syndrome in methadone exposed infants is related to maternal vagal tone changes in response to methadone during pregnancy. While previous research has focused on drug abstinent, methadone maintained women, most drug dependent pregnant women are poly-substance abusers who also use prescription psychiatric medications, alcohol and nicotine. This protocol seeks to further our understanding of the effects of multiple drugs on the fetus, including the co-variate effects of maternal psychological status. Infant neurobehavior and vagal tone will also be evaluated. This research will extend our knowledge of fetal neurobehavioral development and neonatal abstinence syndrome in a realistic population of poly-drug dependent women, potentially altering the way in which these women are evaluated and their infants monitored and treated for neonatal abstinence syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-41
* Single intrauterine fetus
* Free of significant maternal or fetal significant health complications

Exclusion Criteria:

* Development of significant maternal or fetal health complications
* Significant maternal psychopathology that would preclude informed consent
* Unwilling or unable to receive methadone at prescribed times

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Poly drug dependent pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
fetal heart rate | 120 minutes
fetal movement | 120 minutes

SECONDARY OUTCOMES:
neonatal abstinence syndrome | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Addiction and Pregnancy, Baltimore, Maryland, United States

REFERENCES:
- [Result] Jansson LM, Di Pietro JA, Elko A, Williams EL, Milio L, Velez M. Pregnancies exposed to methadone, methadone and other illicit substances, and poly-drugs without methadone: a comparison of fetal neurobehaviors and infant outcomes. Drug Alcohol Depend. 2012 May 1;122(3):213-9. doi: 10.1016/j.drugalcdep.2011.10.003. Epub 2011 Oct 29. PMID 22041255